CLINICAL TRIAL: NCT03824197
Title: Extra-virgin Olive Oil Prevents Mild Cognitive Impairment Conversion to Alzheimer's Disease
Brief Title: Auburn University Research on Olive Oil for Alzheimer's Disease (AU-ROOAD)
Acronym: (AU-ROOAD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Amal Kaddoumi, Professor, Auburn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18-446 MR 1901
Record Dates: First submitted 2019-01-28; First posted 2019-01-31 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Alzheimer Disease; Cerebral Amyloid Angiopathy
MeSH Terms: conditions — Alzheimer Disease; Cerebral Amyloid Angiopathy | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EVOO-phenol high (Other): Extra-virgin olive oil rich with oleocanthal and other phenolic compounds that will be added to daily diet
  Interventions: Other: EVOO
- OO-phenol low (Other): Olive oil with low phenolic content that will be added to daily diet
  Interventions: Other: OO

INTERVENTIONS:
Other: EVOO — Extra-virgin olive oil that is rich with oleocanthal and other phenols.
  Other Names: OC-rich EVOO
  Arms: EVOO-phenol high
Other: OO — Olive oil low in oleocanthal and other phenols.
  Other Names: Olive oil
  Arms: OO-phenol low

SUMMARY:
Until now there is no medical treatment and/or intervention that can slow, stop or reverse the underlying neurodegenerative of Alzheimer's disease (AD). The goal of this study is to demonstrate "Oleocanthal rich-extra-virgin olive oil (EVOO) consumption stops or delay mild cognitive impairment conversion to AD by restoring the blood-brain barrier (BBB) function in humans".

Specific Aims:

1. Evaluate effect of EVOO on the brain function by functional MRI (fMRI) imaging, and BBB function by dynamic contrast-enhanced MRI (DCE-MRI).
2. Evaluate effect of EVOO on cognitive function and on selected biomarkers

ELIGIBILITY:
Inclusion Criteria:

Men and women, experiencing mild cognitive impairment with:

1. Mini-Mental State Exam (MMSE) scores between 18-30 (based on education level
2. memory complaint, have objective memory loss measured by education adjusted scores on Wechsler Memory Scale Logical Memory VI
3. Clinical Dementia Rating (CDR) score 0.5.

Exclusion Criteria:

1. Subjects with contradictions for MRI include: the presence of metal or electronic devices such as metallic joint prostheses, artificial heart valves, an implantable heart defibrillator, a pacemaker, metal clips, cochlear implants, a bullet, shrapnel or any other type of metal fragment; breathing problems or disorders, claustrophobia, inner ear disorders, vertigo or dizziness, tattoos or permanent makeup that contains metal, and body piercing jewelry that cannot be removed.
2. Subjects will be excluded if they are smokers
3. Subjects who have have clinically important medical or neuropsychiatric comorbidity.
4. Subjects who have renal problems or are allergic to the MRI contrast agent.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Effect of olive oil on the BBB intactness | 6 months
  Will be evaluated by DCE-MRI
Effect of olive oil on the brain activity | 6 months
  Will be evaluated by fMRI

SECONDARY OUTCOMES:
Cognitive function | 6 months
  A battery of cognitive tasks to assess memory

CONTACTS AND LOCATIONS:
Overall Officials: Amal Kaddoumi, PhD, Principal Investigator — Auburn University
Locations (1):
- Auburn University, Auburn, Alabama, United States